CLINICAL TRIAL: NCT02619422
Title: Multicenter, Prospective, Randomized, Open, Blinded for the End Point Evaluator to Compare Compliance to Secondary Prevention Measures After Acute Coronary Syndrome and Intensive Cardiac Rehabilitation Program vs Standard Program
Brief Title: More Intensive Cardiac Rehabilitation Programs in Less Time
Acronym: másPORmenos
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Almudena Castro Conde (Other)
Responsible Party: Sponsor-Investigator, Almudena Castro Conde, MD, PhD, Cardiology Department Staff, Hospital Universitario La Paz , Madrid, Spanish Society of Cardiology
Organization: Spanish Society of Cardiology (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: másPORmenos
Record Dates: First submitted 2015-10-04; First posted 2015-12-02 (Estimated); Last update posted 2018-06-06 (Actual); Status verified 2018-06

CONDITIONS: Acute Coronary Syndrome
Keywords: Cardiac rehabilitation programs; Adherence to secondary preventive measures; Acute coronary syndrome; More intensive cardiac rehabilitation program in less time
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intensivo (Other): intensive cardiac rehabilitation program in less time
  Interventions: Other: Intensive cardiac rehabilitation program in less time
- Convencional (No Intervention): standard cardiac rehabilitation program

INTERVENTIONS:
Other: Intensive cardiac rehabilitation program in less time — 2 weeks, 5 days a week, and reinforcement sessions at 3, 6 and 9 months
  Arms: Intensivo

SUMMARY:
To determine if an intensive cardiac rehabilitation program with periodic reinforcements improve the compliance/adherence to secondary preventive measures (physical exercise, mediterranean diet, tobacco abstinence, pharmacological treatment) after an acute coronary syndrome with or without ST segment elevation versus an standard cardiac rehabilitation program

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Equal or older 18 years old
* Acute coronary syndrome with or without ST elevation within last two months
* Being able to do physical exercise
* Being able to understand the educative sessions
* Being able to understand patient information in the consent form

Exclusion Criteria:

* Hemodynamic instability
* Left ventricular ejection fraction (LVEF) < or = 35%
* Heart failure class III -IV (New York Heart Association (NYHA) Functional Classification)
* Refractory angina
* Any pathology for which physical exercise is not indicated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 509 (Actual)
Dates: Start 2015-10; Primary Completion 2018-02 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
Adherence to physical exercise | baseline-12 months
  Assessed in Metabolic Equivalents of Task (METS) from baseline by ergometry
Adherence to Mediterranean diet | baseline-12 months
  Assessed by Mediterranean diet adherence questionnaire (Modified Trichopoulou A,)
Tabacco abstinence | baseline-12 months
  Assessed by cooximetry (less dan 10 ppm)
Number of participants reporting compliance with prescribed treatments | baseline-12 months
  Patient-reported answers form the investigator

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario La Paz, Madrid, Spain

REFERENCES:
- [Derived] Castro-Conde A, Abeytua M, Arrarte Esteban VI, Caravaca Perez P, Dalmau Gonzalez-Gallarza R, Garza Benito F, Hidalgo Urbano RJ, Torres Marques J, Vidal-Perez R, Nunez-Gil IJ. Feasibility and results of an intensive cardiac rehabilitation program. Insights from the MxM (Mas por Menos) randomized trial. Rev Esp Cardiol (Engl Ed). 2021 Jun;74(6):518-525. doi: 10.1016/j.rec.2020.03.029. Epub 2020 Aug 15. English, Spanish. PMID 32807709